CLINICAL TRIAL: NCT07256262
Title: Effect of Functional Magnetic Therapy on Constipation Predominant- Irritable Bowel Syndrome (IBS-C)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Amira Ali Gaber Ali, Principal Investigator, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FPTBSUREC/0204/2225
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional magnetic stimulation (FMS) + Conventional pharmacological therapy (Experimental): It will receive Trans-abdominal FMS plus the conventional pharmacological therapy for 8 weeks.
  Interventions: Device: Functional magnetic stimulation (FMS); Drug: Conventional pharmacological therapy
- Conventional pharmacological therapy (Other): It will receive the conventional pharmacological therapy for 8 weeks.
  Interventions: Drug: Conventional pharmacological therapy

INTERVENTIONS:
Device: Functional magnetic stimulation (FMS) — Every patient will receive 20-minute FMS sessions on the TESLA FORMER device. Each treatment session will consist of one cycle (20 minutes each) based on the treatment area's size and the investigator's discretion. Treatment will be administered by a single applicator secured directly over the abdominal muscles. The device's output intensity will be escalated to a tolerable level depending on patient feedback, with average maximum intensities ranging from 98% to 100% across treatment sessions. The treatment will be 20 minutes long, with several steps including different frequency modulations to achieve stimulation of different muscle fibres.
  Arms: Functional magnetic stimulation (FMS) + Conventional pharmacological therapy
Drug: Conventional pharmacological therapy — Every patient in both groups will receive conventional pharmacological therapy for 8 weeks.

SUMMARY:
The aim of this study is to evaluate the potential benefits of functional magnetic therapy on constipation improvement and related symptoms in patients with IBS-C, including abdominal pain, bloating, bowel habits, and quality of life, as well as to assess patient satisfaction and experience with the therapy.

DETAILED DESCRIPTION:
Functional magnetic stimulation (FMS) has emerged as a promising non-invasive therapeutic approach for managing irritable bowel syndrome (IBS) with predominant constipation, operating through the application of electromagnetic fields that induce electrical currents to modulate neural activity and gastrointestinal function.

Previous research has demonstrated multiple therapeutic benefits of FMS including enhanced bowel motility, increased rectal pain thresholds leading to reduced abdominal pain, improved visceral hypersensitivity, and alleviation of associated psychological symptoms such as anxiety and depression in patients with functional bowel disorders.

The TESLA Former is a high-intensity Functional Magnetic Stimulation (FMS) device, that operates through multiple therapeutic mechanisms in treating IBS with predominant constipation: it delivers electromagnetic pulses to strengthen pelvic floor muscles and enhance defecation dynamics while modulating the brain-gut axis through stimulation of pudendal and sacral nerves (S2-S4); additionally, it influences the enteric nervous system (ENS) to normalize gut peristalsis and bowel transit, while simultaneously reducing inflammation and stress response through autonomic nervous system modulation, ultimately addressing both the physical and psychological components of IBS by improving muscle coordination, reducing visceral hypersensitivity, and promoting a balanced gut microbiota environment.

Research has demonstrated that the TESLA Former delivers significant therapeutic outcomes in treating IBS, including improved bowel function with increased frequency and ease of bowel movements, reduced abdominal discomfort manifested through diminished bloating and visceral pain, and enhanced quality of life (QOL) through reduced laxative dependency and improved symptom control; notably, this non-invasive therapy demonstrates excellent safety and tolerability profile.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of IBS-C based on Rome IV criteria.
2. Age: Adults aged 18-65 years.
3. Symptom Duration: Symptoms present for at least 6 months before diagnosis.
4. Ability to Consent: Patients must be able to provide informed consent and comply with study requirements.

Exclusion Criteria:

1. Presence of Alarm Features or Red Flags:

   * Unexplained weight loss.
   * Blood in stool or rectal bleeding.
   * Anaemia (iron deficiency anaemia).
   * Persistent vomiting.
2. Underlying Organic Diseases:

   - Conditions such as inflammatory bowel disease (IBD), celiac disease, colorectal cancer, or other structural gastrointestinal abnormalities.
3. Pregnancy or Lactation.
4. Surgery or Anatomic Alterations: History of major gastrointestinal surgeries (e.g., bowel resection) that could affect bowel function.
5. Contraindications to the Procedure:

   * Patients with pacemaker
   * Condition that can compromise increased abdominal pressure, such as hernia.
   * Condition that can prevent adequate performance of abdominal muscle tension.
   * Recent thoracic or abdominal surgery precluding the use of functional magnetic therapy.
   * Rib fractures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-28 (Estimated); Primary Completion 2026-01-28 (Estimated); Study Completion 2026-02-14 (Estimated)

PRIMARY OUTCOMES:
IBS Severity Scoring System (IBS-SSS) | 8 weeks
  It is a tool used to assess the severity of symptoms in patients with irritable bowel syndrome (IBS). It consists of five key questions that measure the intensity and impact of symptoms such as abdominal pain, bloating, bowel movement frequency, and the overall effect of IBS on QOL. Each symptom is rated on a scale from 0 to 100, and the total score ranges from 0 to 500. The total score helps categorize the severity of IBS as mild (75-175), moderate (175-300), or severe (300-500). The IBS-SSS is valuable for clinicians to monitor symptom progression, evaluate treatment effectiveness, and track the impact of IBS on a patient's daily life.
Complete Spontaneous Bowel Movements (CSBMs) | 8 weeks
  A complete spontaneous bowel movement (CSBM) is defined as a natural, voluntary bowel movement without the need for medical intervention, medications, or external aids. It involves the elimination of waste with a feeling of complete evacuation, occurring regularly (from three times a week to three times a day). CSBM typically is accompanied by the sensation of complete emptying and occurs without laxative use in the previous 24 hours, indicating normal gastrointestinal health and function. It is used as a clinical marker to evaluate digestive health, particularly in assessing conditions like irritable bowel syndrome.
Bristol Stool Scale Assessment (BSS) | 8 weeks
  It is a medical tool used to classify stool consistency and type, helping in assessing bowel health. The scale consists of seven types of stool, ranging from Type 1 (hard and lumpy) to Type 7 (liquid and watery). Types 3 and 4 are generally considered normal, with Type 3 resembling a sausage shape with cracks and Type 4 being smooth and soft, similar to a sausage or snake. It helps in monitoring bowel function, determining the effectiveness of treatments, and providing insight into gastrointestinal health.

SECONDARY OUTCOMES:
The Visual Analog Scale (VAS) | 8 weeks
  The VAS consists of a straight line, typically 10 cm in length, where one end represents "no pain" and the other end represents "worst possible pain". Patients will be asked to mark a point on the line that represents the severity of their pain, with the position of the mark indicating their pain level. The scale is then measured in centimetres or millimeters, with higher values indicating more intense pain.
Pain Interference with Activities | 8 weeks
  It refers to the interference of pain with different activities such as walking, sitting, working light or heavy work and It grades from (None □ Mild □ Moderate □ Severe Complete).
Patient Assessment of Constipation Quality of Life (PAC-QOL ) | 8 weeks
  It is a self-reported questionnaire designed to assess the impact of constipation on a patient's quality of life. It helps evaluate the psychological, social, and physical effects of constipation on daily living. The questionnaire consists of a series of statements that the patient rates based on their experiences over the past week, with responses typically ranging from "not at all" to "very much. The PAC-QOL is divided into four domains.

CONTACTS AND LOCATIONS:
Overall Officials: Tamer I Abo Elyazed, PhD, Study Chair — Assistant Professor, Beni-Suef University; Ragaey Ahmad Eid, PhD, Study Director — Assistant Professor, Beni-Suef University; Marwa Mohamed Eleawa, Study Director — Lecturer, Beni-Suef University
Locations (1):
- Beni-Suef University, Banī Suwayf, Egypt